CLINICAL TRIAL: NCT05800184
Title: Finnish Imaging of Shoulder Trauma
Acronym: FIMAGE-T
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Professor Teppo Järvinen, Professor, Helsinki University Central Hospital
Other Study IDs: HUS/13603/2022
Record Dates: First submitted 2023-03-09; First posted 2023-04-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Shoulder Pain; Shoulder Injuries; Rotator Cuff Tears; Glenoid Labrum Tear
Keywords: Shoulder; Injury; Rotator Cuff; Magnetic resonance Imaging
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries; Rotator Cuff Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with a shoulder injury: Individuals from a population based sample of 600 individuals aged 40 to 75 years that sustain a shoulder injury or a sudden onset of significant shoulder symptoms.

SUMMARY:
The FIMAGE-Trauma study is an extension of the FIMAGE study and aims to answer the question if rotator cuff tears found on shoulder imaging after a shoulder injury are caused by the index trauma or are rather incidental findings. Eligible participants of the FIMAGE study will be invited to a follow up visit in the case of a shoulder injury or a sudden onset of significant shoulder symptoms (within a 2-year time frame). These findings will then be compared to the baseline data collected in the FIMAGE study (including the comparison of pre-injury and post-injury MRI:s)

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Participated in the FIMAGE
* Baseline MRI from FIMAGE study available

Exclusion Criteria:

* Contraindications to MRI
* Previous shoulder joint replacement
* Previous rotator cuff surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects from a population based sample (FIMAGE study participants) who sustain a shoulder injury or sudden onset of significant shoulder symptoms within 2 years after the FIMAGE research visit.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rotator Cuff Integrity on Shoulder Magnetic Resonance Imaging (MRI) | At baseline
  Bilateral shoulder MRI comparing the integrity of the rotator cuff tendons on pre-injury and post-injury MRI scans. Each of the four rotator cuff tendons (supraspinatus, infraspinatus, teres minor, subscapularis) will be assessed and graded for structural changes (normal, tendinopathy, partial thickness tear, full thickness tear). The dimensions of full thickness tears will be measured and recorded (size in millimeters).
Shoulder Pain and Disability Index (SPADI) | At baseline
  Patient reported outcome measure. The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. A SPADI total score ranging from 0 (best) to 100 (worst) is produced by averaging the two subscale scores.
Constant -Murley Score | At baseline
  The Constant-Murley Score was designed to assess the functional state of a shoulder and contains both physician- completed and patient-reported portions. The four domains include pain (15 possible points), activities of daily living (20 possible points), mobility (40 possible points), and strength (25 possible points). Scores range from 0 points (most disability) to 100 points (least disability).

SECONDARY OUTCOMES:
Subjective Shoulder Value (SSV) | At baseline
  The SSV score is defined as the subjective evaluation by the patient of shoulder function, expressed as a percentage of a normal shoulder. This score ranges from 0 to 100%.
Pain NRS | At baseline
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".

OTHER OUTCOMES:
Clinical Shoulder Examination | At baseline
  The clinical examination will include orthopaedic shoulder tests used to assess rotator cuff integrity (internal rotation lag sign, lift off, press belly, hornblower sign, bear hug test, drop arm sign, external rotation lag sign).

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No